CLINICAL TRIAL: NCT00435734
Title: Evaluation of the Intervention Program "Obeldicks" for Obese Children and Adolescents
Brief Title: Obesity Intervention "Obeldicks" for Obese Children, Adolescents and Their Parents
Acronym: Obeldicks
Status: Active, not recruiting | Type: Observational
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, Thomas Reinehr, Head of Department of Pediatric Endocrinology Diabetes and Nutrition Medicine, University of Witten/Herdecke
Other Study IDs: GFEL011174506
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — frozen Serum probes

INTERVENTIONS:
Behavioral: obesity intervention

SUMMARY:
The intervention program "Obeldicks" was developed for obese children aged 6 to 16 years. This intervention is gender- and age specific. The 12-months intervention is based on nutrition course, behaviour therapy and exercise therapy. The evaluation compromised quality of structure, process and results of the intervention. Primary outcome measure is change of weight status as standard deviation score of BMI. Furthermore, cardiovascular risk factor profile, hormones (e.g. iGF-I, thyroid hormones, vitamin D status)adipocytokines, GI- hormones, intima media thickness are measured prior to and after the one-year intervention. The changes of these hormones and adipocytokines will allow to answer the questions whether the alterations of these hormones are a cause or consequence of overweight. Additionally, a genetic screening is performed to characterize the participants to probably predict response to intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI> 97. percentile for age and gender

Exclusion Criteria:

* Psychiatric disorders
* Endocrine disorders

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: clinic based study of obese children
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 1999-07; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
change of BMI-SDS | 20 years

SECONDARY OUTCOMES:
change of GI hormones | 10 years
change of adipocytokines | 10 years
change of cardiovascualr risk factors | 10 years
change of metabolomics | 10 years
change of psychological variables | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Reinehr, Principal Investigator — Vestische Children´s Hospital
Locations (1):
- Vestische Children´s Hospital, Datteln, Germany

REFERENCES:
- [Derived] Reinehr T, Kulle A, Barth A, Ackermann J, Lass N, Holterhus PM. Sex Hormone Profile in Pubertal Boys With Gynecomastia and Pseudogynecomastia. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgaa044. doi: 10.1210/clinem/dgaa044. PMID 31996898
- [Derived] Rothermel J, Lass N, Barth A, Reinehr T. Link between omentin-1, obesity and insulin resistance in children: Findings from a longitudinal intervention study. Pediatr Obes. 2020 May;15(5):e12605. doi: 10.1111/ijpo.12605. Epub 2019 Dec 16. PMID 31840425
- [Derived] Reinehr T, Bosse C, Lass N, Rothermel J, Knop C, Roth CL. Effect of Weight Loss on Puberty Onset in Overweight Children. J Pediatr. 2017 May;184:143-150.e1. doi: 10.1016/j.jpeds.2017.01.066. Epub 2017 Feb 24. PMID 28238482
- [Derived] Reinehr T, Lass N, Toschke C, Rothermel J, Lanzinger S, Holl RW. Which Amount of BMI-SDS Reduction Is Necessary to Improve Cardiovascular Risk Factors in Overweight Children? J Clin Endocrinol Metab. 2016 Aug;101(8):3171-9. doi: 10.1210/jc.2016-1885. Epub 2016 Jun 10. PMID 27285295
- [Derived] Hellmuth C, Kirchberg FF, Lass N, Harder U, Peissner W, Koletzko B, Reinehr T. Tyrosine Is Associated with Insulin Resistance in Longitudinal Metabolomic Profiling of Obese Children. J Diabetes Res. 2016;2016:2108909. doi: 10.1155/2016/2108909. Epub 2015 Dec 21. PMID 26881241
- [Derived] Reinehr T, Elfers C, Lass N, Roth CL. Irisin and its relation to insulin resistance and puberty in obese children: a longitudinal analysis. J Clin Endocrinol Metab. 2015 May;100(5):2123-30. doi: 10.1210/jc.2015-1208. Epub 2015 Mar 17. PMID 25781361
- [Derived] Reinehr T, Wolters B, Knop C, Lass N, Holl RW. Strong effect of pubertal status on metabolic health in obese children: a longitudinal study. J Clin Endocrinol Metab. 2015 Jan;100(1):301-8. doi: 10.1210/jc.2014-2674. PMID 25243573
- [Derived] Reinehr T, Wolters B, Roth CL, Hinney A. FTO gene: association to weight regain after lifestyle intervention in overweight children. Horm Res Paediatr. 2014;81(6):391-6. doi: 10.1159/000358328. Epub 2014 May 7. PMID 24819256
- [Derived] Reinehr T, Kulle A, Wolters B, Knop C, Lass N, Welzel M, Holterhus PM. Relationships between 24-hour urinary free cortisol concentrations and metabolic syndrome in obese children. J Clin Endocrinol Metab. 2014 Jul;99(7):2391-9. doi: 10.1210/jc.2013-4398. Epub 2014 Mar 26. PMID 24670085
- [Derived] Roth CL, Hinney A, Schur EA, Elfers CT, Reinehr T. Association analyses for dopamine receptor gene polymorphisms and weight status in a longitudinal analysis in obese children before and after lifestyle intervention. BMC Pediatr. 2013 Nov 27;13:197. doi: 10.1186/1471-2431-13-197. PMID 24283216
- [Derived] Uysal Y, Wolters B, Knop C, Reinehr T. Components of the metabolic syndrome are negative predictors of weight loss in obese children with lifestyle intervention. Clin Nutr. 2014 Aug;33(4):620-5. doi: 10.1016/j.clnu.2013.09.007. Epub 2013 Sep 18. PMID 24075648
- [Derived] Reinehr T, Kulle A, Wolters B, Lass N, Welzel M, Riepe F, Holterhus PM. Steroid hormone profiles in prepubertal obese children before and after weight loss. J Clin Endocrinol Metab. 2013 Jun;98(6):E1022-30. doi: 10.1210/jc.2013-1173. Epub 2013 May 23. PMID 23703723
- [Derived] Volckmar AL, Putter C, Song JY, Graniger J, Knoll N, Wolters B, Hebebrand J, Scherag A, Reinehr T, Hinney A. Analyses of non-synonymous obesity risk alleles in SH2B1 (rs7498665) and APOB48R (rs180743) in obese children and adolescents undergoing a 1-year lifestyle intervention. Exp Clin Endocrinol Diabetes. 2013 Jun;121(6):334-7. doi: 10.1055/s-0033-1334875. Epub 2013 Mar 21. PMID 23519644
- [Derived] Reinehr T, Wunsch R, Putter C, Scherag A. Relationship between carotid intima-media thickness and metabolic syndrome in adolescents. J Pediatr. 2013 Aug;163(2):327-32. doi: 10.1016/j.jpeds.2013.01.032. Epub 2013 Feb 26. PMID 23485031
- [Derived] Wolters B, Lass N, Reinehr T. TSH and free triiodothyronine concentrations are associated with weight loss in a lifestyle intervention and weight regain afterwards in obese children. Eur J Endocrinol. 2013 Feb 15;168(3):323-9. doi: 10.1530/EJE-12-0981. Print 2013 Mar. PMID 23211576
- [Derived] Reinehr T, Woelfle J, Wunsch R, Roth CL. Fibroblast growth factor 21 (FGF-21) and its relation to obesity, metabolic syndrome, and nonalcoholic fatty liver in children: a longitudinal analysis. J Clin Endocrinol Metab. 2012 Jun;97(6):2143-50. doi: 10.1210/jc.2012-1221. Epub 2012 Mar 21. PMID 22438225
- [Derived] Scherag A, Kleber M, Boes T, Kolbe AL, Ruth A, Grallert H, Illig T, Heid IM, Toschke AM, Grau K; NUGENOB Consortium; Sorensen TI, Hebebrand J, Hinney A, Reinehr T. SDCCAG8 obesity alleles and reduced weight loss after a lifestyle intervention in overweight children and adolescents. Obesity (Silver Spring). 2012 Feb;20(2):466-70. doi: 10.1038/oby.2011.339. Epub 2011 Nov 17. PMID 22095114
- [Derived] Knoll N, Volckmar AL, Putter C, Scherag A, Kleber M, Hebebrand J, Hinney A, Reinehr T. The fatty acid amide hydrolase (FAAH) gene variant rs324420 AA/AC is not associated with weight loss in a 1-year lifestyle intervention for obese children and adolescents. Horm Metab Res. 2012 Jan;44(1):75-7. doi: 10.1055/s-0031-1291306. Epub 2011 Nov 8. PMID 22068813
- [Derived] Lass N, Kleber M, Winkel K, Wunsch R, Reinehr T. Effect of lifestyle intervention on features of polycystic ovarian syndrome, metabolic syndrome, and intima-media thickness in obese adolescent girls. J Clin Endocrinol Metab. 2011 Nov;96(11):3533-40. doi: 10.1210/jc.2011-1609. Epub 2011 Aug 31. PMID 21880803
- [Derived] Kleber M, Schwarz A, Reinehr T. Obesity in children and adolescents: relationship to growth, pubarche, menarche, and voice break. J Pediatr Endocrinol Metab. 2011;24(3-4):125-30. doi: 10.1515/jpem.2011.089. PMID 21648278
- [Derived] Reinehr T, Woelfle J, Roth CL. Lack of association between apelin, insulin resistance, cardiovascular risk factors, and obesity in children: a longitudinal analysis. Metabolism. 2011 Sep;60(9):1349-54. doi: 10.1016/j.metabol.2011.02.005. Epub 2011 Apr 12. PMID 21489579
- [Derived] Vogel CI, Boes T, Reinehr T, Roth CL, Scherag S, Scherag A, Hebebrand J, Hinney A. Common variants near MC4R: exploring gender effects in overweight and obese children and adolescents participating in a lifestyle intervention. Obes Facts. 2011;4(1):67-75. doi: 10.1159/000324557. Epub 2011 Feb 22. PMID 21372613
- [Derived] Reinehr T, Scherag A, Wang HJ, Roth CL, Kleber M, Scherag S, Boes T, Vogel C, Hebebrand J, Hinney A. Relationship between MTNR1B (melatonin receptor 1B gene) polymorphism rs10830963 and glucose levels in overweight children and adolescents. Pediatr Diabetes. 2011 Jun;12(4 Pt 2):435-41. doi: 10.1111/j.1399-5448.2010.00738.x. Epub 2011 Mar 3. PMID 21366812
- [Derived] Reinehr T, Kleber M, Toschke AM, Woelfle J, Roth CL. Longitudinal association between IGFBP-1 levels and parameters of the metabolic syndrome in obese children before and after weight loss. Int J Pediatr Obes. 2011 Aug;6(3-4):236-43. doi: 10.3109/17477166.2010.544739. Epub 2011 Jan 3. PMID 21198359
- [Derived] Kleber M, deSousa G, Papcke S, Wabitsch M, Reinehr T. Impaired glucose tolerance in obese white children and adolescents: three to five year follow-up in untreated patients. Exp Clin Endocrinol Diabetes. 2011 Mar;119(3):172-6. doi: 10.1055/s-0030-1263150. Epub 2010 Sep 8. PMID 20827664
- [Derived] Kleber M, Lass N, Papcke S, Wabitsch M, Reinehr T. One-year follow-up of untreated obese white children and adolescents with impaired glucose tolerance: high conversion rate to normal glucose tolerance. Diabet Med. 2010 May;27(5):516-21. doi: 10.1111/j.1464-5491.2010.02991.x. PMID 20536946
- [Derived] Reinehr T, Roth CL, Enriori PJ, Masur K. Changes of dipeptidyl peptidase IV (DPP-IV) in obese children with weight loss: relationships to peptide YY, pancreatic peptide, and insulin sensitivity. J Pediatr Endocrinol Metab. 2010 Jan-Feb;23(1-2):101-8. doi: 10.1515/jpem.2010.23.1-2.101. PMID 20432813
- [Derived] Reinehr T, Kleber M, Lass N, Toschke AM. Body mass index patterns over 5 y in obese children motivated to participate in a 1-y lifestyle intervention: age as a predictor of long-term success. Am J Clin Nutr. 2010 May;91(5):1165-71. doi: 10.3945/ajcn.2009.28705. Epub 2010 Mar 10. PMID 20219965
- [Derived] Reinehr T, Kleber M, Toschke AM. Former small for gestational age (SGA) status is associated to changes of insulin resistance in obese children during weight loss. Pediatr Diabetes. 2010 Sep;11(6):431-7. doi: 10.1111/j.1399-5448.2009.00624.x. Epub 2009 Dec 30. PMID 20051022
- [Derived] Reinehr T, Kleber M, de Sousa G, Andler W. Leptin concentrations are a predictor of overweight reduction in a lifestyle intervention. Int J Pediatr Obes. 2009;4(4):215-23. doi: 10.3109/17477160902952464. PMID 19922035
- [Derived] Roth CL, Enriori PJ, Gebhardt U, Hinney A, Muller HL, Hebebrand J, Reinehr T, Cowley MA. Changes of peripheral alpha-melanocyte-stimulating hormone in childhood obesity. Metabolism. 2010 Feb;59(2):186-94. doi: 10.1016/j.metabol.2009.06.031. Epub 2009 Sep 18. PMID 19766264
- [Derived] Reinehr T, Wunsch R. Relationships between cardiovascular risk profile, ultrasonographic measurement of intra-abdominal adipose tissue, and waist circumference in obese children. Clin Nutr. 2010 Feb;29(1):24-30. doi: 10.1016/j.clnu.2009.06.004. Epub 2009 Jul 2. PMID 19576664
- [Derived] Reinehr T, Panteliadou A, de Sousa G, Andler W. Insulin-like growth factor-I, insulin-like growth factor binding protein-3 and growth in obese children before and after reduction of overweight. J Pediatr Endocrinol Metab. 2009 Mar;22(3):225-33. doi: 10.1515/jpem.2009.22.3.225. PMID 19492578
- [Derived] Reinehr T, Kleber M, Toschke AM. Lifestyle intervention in obese children is associated with a decrease of the metabolic syndrome prevalence. Atherosclerosis. 2009 Nov;207(1):174-80. doi: 10.1016/j.atherosclerosis.2009.03.041. Epub 2009 Apr 5. PMID 19442975
- [Derived] Reinehr T, Schmidt C, de Sousa G, Andler W. Association between leptin and transaminases: 1-year follow-up study in 180 overweight children. Metabolism. 2009 Apr;58(4):497-503. doi: 10.1016/j.metabol.2008.11.007. PMID 19303970
- [Derived] Reinehr T, Schmidt C, Toschke AM, Andler W. Lifestyle intervention in obese children with non-alcoholic fatty liver disease: 2-year follow-up study. Arch Dis Child. 2009 Jun;94(6):437-42. doi: 10.1136/adc.2008.143594. Epub 2009 Feb 17. PMID 19224892
- [Derived] Reinehr T, Kleber M, Toschke AM. Small for gestational age status is associated with metabolic syndrome in overweight children. Eur J Endocrinol. 2009 Apr;160(4):579-84. doi: 10.1530/EJE-08-0914. Epub 2009 Jan 20. PMID 19155319
- [Derived] Muller TD, Hinney A, Scherag A, Nguyen TT, Schreiner F, Schafer H, Hebebrand J, Roth CL, Reinehr T. 'Fat mass and obesity associated' gene (FTO): no significant association of variant rs9939609 with weight loss in a lifestyle intervention and lipid metabolism markers in German obese children and adolescents. BMC Med Genet. 2008 Sep 17;9:85. doi: 10.1186/1471-2350-9-85. PMID 18799002
- [Derived] Reinehr T, Roth CL. Fetuin-A and its relation to metabolic syndrome and fatty liver disease in obese children before and after weight loss. J Clin Endocrinol Metab. 2008 Nov;93(11):4479-85. doi: 10.1210/jc.2008-1505. Epub 2008 Aug 26. PMID 18728159
- [Derived] Reinehr T, Stoffel-Wagner B, Roth CL. Retinol-binding protein 4 and its relation to insulin resistance in obese children before and after weight loss. J Clin Endocrinol Metab. 2008 Jun;93(6):2287-93. doi: 10.1210/jc.2007-2745. Epub 2008 Apr 8. PMID 18397979
- [Derived] Reinehr T, Wunsch R, de Sousa G, Toschke AM. Relationship between metabolic syndrome definitions for children and adolescents and intima-media thickness. Atherosclerosis. 2008 Jul;199(1):193-200. doi: 10.1016/j.atherosclerosis.2007.09.041. Epub 2007 Nov 26. PMID 18031749
- [Derived] Reinehr T, de Sousa G, Roth CL. Obestatin and ghrelin levels in obese children and adolescents before and after reduction of overweight. Clin Endocrinol (Oxf). 2008 Feb;68(2):304-10. doi: 10.1111/j.1365-2265.2007.03042.x. Epub 2007 Sep 14. PMID 17854392
- [Derived] Reinehr T, de Sousa G, Alexy U, Kersting M, Andler W. Vitamin D status and parathyroid hormone in obese children before and after weight loss. Eur J Endocrinol. 2007 Aug;157(2):225-32. doi: 10.1530/EJE-07-0188. PMID 17656603